CLINICAL TRIAL: NCT00311415
Title: A Phase III, Multi-Center, Open-Label, Controlled, Randomized Study to Evaluate the Immunogenicity, Safety, Tolerability and the Ability to Prime for Memory of Chiron Meningococcal C Conjugate Vaccine When Administered to Healthy Infants as One Dose Given at 2 or 6 Months of Age With a Booster at 12-16 Months of Age, in Comparison to Two Doses in the First Year of Life, Given Two Months Apart, With a Booster at 12-16 Months of Age; and in Comparison to One Dose Given at 12-16 Months of Age
Brief Title: Immunogenicity, Safety, Tolerability and Ability to Prime for Memory of Meningococcal C Conjugate Vaccine in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M14P6; Impact N° 919
Record Dates: First submitted 2006-04-03; First posted 2006-04-06 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Prevention of Meningococcal Infection
Keywords: Prevention of Meningococcal Meningitis; meningococcal vaccines; conjugate; immunology; infant; antibody persistence
MeSH Terms: interventions — serogroup C meningococcal conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: 2+4 Months (2-doses) (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 2: 2 Months (1-dose) (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 3: 6 Months (1-dose) (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 4: 12-16 Months (1 dose in the second year of life) (Active Comparator)
  Interventions: Biological: Meningococcal C conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C conjugate vaccine — Meningococcal conjugate vaccine, active comparator.
  Groups 1 to 3 were given a booster dose in the second year of life at 12-16 months of age

SUMMARY:
Immunogenicity, Safety, Tolerability and Ability to Prime for Memory of Meningococcal C Conjugate Vaccine in healthy children

DETAILED DESCRIPTION:
The aim of this study is to investigate the immunogenicity offered by MenCC vaccine when administered in different schedules at different years of life: 2 doses in the first year of life given 2 months apart (at 2 and 4 months of age), with a booster in the second year of life, or 1 dose in the first year of life (at 2 or 6 months of age), with a booster in the second year of life, or only 1 dose in the second year of life.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants

Exclusion Criteria:

* known hypersensitivity to any vaccine component
* significant acute or chronic infections
* previously ascertained or suspected disease caused by N. meningitidis
* previous household contact with an individual with a positive culture of N. meningitidis serogroup C

Ages: 7 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 257 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Demonstration of non-inferiority of memory antibody response after 1 dose of MenC Vaccine administered to healthy infants at 2 to 6 months of age and as first, second or third dose in the second year of life,as measured by rBCA. | Overall study period

SECONDARY OUTCOMES:
Evaluation and comparison of antibody response and its persistence in terms of GMT and percent responders, as measured by rBCA. | Overall study period

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (2):
- Mainz, Kehl, Neumünster, Ettenheim, Germany
- Kraków, Lubartów, Lublin, Bydgosczcz, Poland